CLINICAL TRIAL: NCT02211040
Title: Effect Evaluation of an eHealth Intervention to Promote Self-regulation of Physical Activity and Fruit and Vegetable Intake Among Adults in General Practice
Brief Title: eHealth Intervention to Promote Self-regulation of Physical Activity and Fruit and Vegetable Intake Among Adults Who Visit General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Welfare, Public Health and Family, Flemish government, Belgium (Unknown)
Responsible Party: Principal Investigator, Vakgroepsport, Professor doctor Ilse De Bourdeaudhuij, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BE670201421382
Record Dates: First submitted 2014-07-18; First posted 2014-08-07 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Physical Activity; Fruit and Vegetable Intake; Self-regulation; Empowerment
Keywords: Intervention Mapping Protocol; physical activity; fruit intake; vegetable intake; computer tailoring; eHealth; self-regulation; goal setting; problem solving; general practice
MeSH Terms: conditions — Motor Activity; Self-Control; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No general practitioner involvement (Experimental): The selection and motivation of adults will be conducted by a researcher in the waiting room. There is no extra motivation of the general practitioner.
  Interventions: Behavioral: My Plan
- General practitioner involvement (Experimental): An intervention group in which general practitioners select and motivate adults to be more physical active and eat more fruit and vegetables.
  Interventions: Behavioral: My Plan

INTERVENTIONS:
Behavioral: My Plan — The intervention consists of three sessions for each behaviour (ie., physical activity, fruit and vegetables intake) and is available on a website and tablets to deliver it in general practice.
  Adults can start session one on a tablet in general practice or on their own computer at home, after receiving a flyer in general practice.
  In this first session adults receive general information, monitor their behaviour and receive tailored feedback to increase awareness.
  Adults are also guided to set goals and self-efficacy is increased by modeling and problem solving methods.
  In the second and third session, adults can evaluate if they reached their goals, make coping plans and adapt their action plans.

SUMMARY:
The investigators have developed an eHealth intervention based on self-regulation for the promotion of self-regulation of physical activity and fruit and vegetable intake among adults who visit general practice. Effectiveness of the intervention will be evaluated in a three-arm clustered quasi-experimental design in general practice.

DETAILED DESCRIPTION:
To increase effect sizes and reach of computer tailored interventions, the theory of self-regulation was used, motivational and volitional determinants were targeted and the intervention was not served as a stand-alone intervention but was delivered in general practice. The intervention consists of three sessions for each behaviour (ie., physical activity, fruit and vegetables intake) and is available on a website and tablets to deliver it in general practice. Adults can start session one on a tablet in general practice or on their own computer at home, after receiving a flyer in general practice. In this first session adults receive general information, monitor their behaviour and receive tailored feedback to increase awareness. Adults are also guided to set goals and self-efficacy is increased by modeling and problem solving methods. In the second and third session, adults can evaluate if they reached their goals, make coping plans and adapt their action plans. To ensure the feasibility of implementing the intervention in general practice, general practitioners were involved from the beginning of the development.

A three-arm clustered quasi-experimental design will be used to evaluate the effectiveness of the intervention. Therefore, general practitioners will be recruited and patients will be randomly assigned at general practice level. Within each practice, patients can be allocated in three groups. Group one is an intervention group in which general practitioners select and motivate adults to use the intervention. In group two, the selection and motivation of adults will be conducted by a researcher in the waiting room and finally, group three will be a control group in which adults are also selected by a researcher. The distinction between the two intervention groups is made to evaluate if general practitioners influence when recruiting participants leads to beneficial effects compared to when investigators recruit participants. Furthermore, it will also be investigated if the implementation of the intervention by general practitioners is feasible.

In the intervention groups, adults are asked to complete session one (S1) and measurements questions on a tablet in general practice or are referred with a flyer to do this at their computer at home. Adults, who do not use the tablet, have to fill in a short questionnaire and leave their email address to send them a reminder email to complete session one at home. In session one, adults choose themselves for which behaviour(s) they want to complete the intervention. One week (S2) and one month (S3) after session one is completed, adults will receive an email to respectively start session two and three for the chosen behaviour(s). In the control group, adults have to fill in a questionnaire at base line in general practice or at home (C1) and one month post intervention (C2).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Having access to internet

Exclusion Criteria:

* No access to internet
* Younger than 18 years
* Not understanding the Dutch Language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
"Change from Baseline in physical activity level at 1 and 6 months" | After 1 and 6 months
  Amount of physical activity per day and per week
"Change from Baseline in fruit and vegetable intake at 1 and 6 months" | After 1 and 6 months

SECONDARY OUTCOMES:
"Change from Baseline in scores on self-regulation skills at 1 and 6 months" | After 1 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jolien Plaete, Ghent, East Flanders, Belgium

REFERENCES:
- [Derived] Van Dyck D, Plaete J, Cardon G, Crombez G, De Bourdeaudhuij I. Effectiveness of the self-regulation eHealth intervention 'MyPlan1.0.' on physical activity levels of recently retired Belgian adults: a randomized controlled trial. Health Educ Res. 2016 Oct;31(5):653-64. doi: 10.1093/her/cyw036. Epub 2016 Jul 15. PMID 27422898
- [Derived] Plaete J, Crombez G, Van der Mispel C, Verloigne M, Van Stappen V, De Bourdeaudhuij I. Effect of the Web-Based Intervention MyPlan 1.0 on Self-Reported Fruit and Vegetable Intake in Adults Who Visit General Practice: A Quasi-Experimental Trial. J Med Internet Res. 2016 Feb 29;18(2):e47. doi: 10.2196/jmir.5252. PMID 26929095
- See also: Funding — https://steunpuntwvg.be/